CLINICAL TRIAL: NCT04445675
Title: Investigation of the Effect of Support Provided for Breastfeeding and the Feeding of Infants' With Breast Milk on Hospitalization Due to Jaundice
Brief Title: The Effect of Breastfeeding Support on Hospitalization Due to Jaundice
Acronym: Breastfeeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Özge Karakaya Suzan, reseaech asistant, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ozge
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Hyperbilirubinemia, Neonatal; Jaundice, Neonatal
Keywords: Newborn; Hyperbilirubinemia; Breastfeeding support; Nurse
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Jaundice, Neonatal; Hyperbilirubinemia | interventions — Palliative Care; Lactation; Milk, Human

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Single-blind (researchers are not blind) randomization will be provided since the mothers will be provided with support for breastfeeding and the feeding of infants' with breast milk by the researchers. The statistician was also blinded for the data analysis purpose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The support for breastfeeding and the feeding of infants' with breast milk will be conducted in one stage for the experimental group. (1) breastfeeding support education. The content of the support for breastfeeding and the feeding of infants' with breast milk and the materials used were determined by the researchers in accordance with the literature. The content of the support for breastfeeding and the feeding of infants' with breast milk consists of the titles of the importance of breastfeeding and breast milk, the effect of breast milk on preventing jaundice, the importance of early start of breastfeeding, breastfeeding techniques and positions in infants, milking, storage and later use of milk, increasing the quantity and quality of milk, and nutrition of the mother during breastfeeding. Breastfeeding support will be provided in the postpartum service and lactation outpatient clinic of the relevant hospital.
  Interventions: Other: Support for breastfeeding and the feeding of infants' with breast milk
- Control Groups (No Intervention): The infants in the control group will be followed up in routine service. No intervention will be made.

INTERVENTIONS:
Other: Support for breastfeeding and the feeding of infants' with breast milk — The content of the support for breastfeeding and the feeding of infants' with breast milk consists of the titles of the importance of breastfeeding and breast milk, the effect of breast milk on preventing jaundice, the importance of early start of breastfeeding, breastfeeding techniques and positions in infants, milking, storage and later use of milk, increasing the quantity and quality of milk, and nutrition of the mother during breastfeeding.
  Arms: Experimental

SUMMARY:
Neonatal jaundice is the most common reason for rehospitalization after postnatal discharge. Jaundice due to breastfeeding failure is an important subtype of pathological neonatal jaundice. Typically, it occurs with lactation failure, which results in dehydration (reducing urine output), significant weight loss (>10% of birth weight) and sometimes hypernatremia, during the first postnatal week. Jaundice caused by breastfeeding failure is observed in one third (31.8%) of total cases of pathological neonatal jaundice requiring rehospitalization. Jaundice lasts for an average of 6.8 days and the length of hospital stay takes up to 3 days. Jaundice due to breastfeeding failure requires focused efforts for a program structured with breastfeeding education and special breastfeeding support. This support causes the role of nurses to become even more important. The aim of this study is to investigate the effect of support provided for breastfeeding and the feeding of infants' with breast milk on hospitalization due to jaundice.

Research Hypotheses:

H0: The support provided for breastfeeding and the feeding of infants' with breast milk has no effect on hospitalization due to jaundice.

H1: The support provided for breastfeeding and the feeding of infants' with breast milk affects the consequences of hospitalization due to jaundice.

DETAILED DESCRIPTION:
Background: Neonatal jaundice is a condition that is accompanied by hyperbilirubinemia. Almost all newborns (60% term and 80% preterm) have more than 5mg/dl of bilirubin during the first week of life, and approximately 6% of term infants may have levels exceeding 15 mg/dl (Young Infants Clinical Signs Study Group, 2008). It is one of the most common causes of morbidity during the first week of life. High serum bilirubin level leads to serious consequences and neurologic disorders in some of the infants with jaundice. 5-10% of these newborns have clinically important neonatal jaundice that requires treatment and care to prevent neurotoxicity and reduce serum bilirubin level (Madan, Mac Mohan, Stevenson, 2005). Recent studies in the literature have shown that there is a strong relationship between hyperbilirubinemia and breastfeeding (Garg, 2018; Flaherman 2017). In a study, it was indicated that breastfed infants had lower bilirubin levels on postnatal day 3 compared to infants fed with infant formula. The problem of jaundice that increases due to insufficient intake of breast milk/breastfeeding is usually underestimated, an exaggerated physiological jaundice treatment is often administered (symptomatically phototherapy), and breastfeeding problems are neglected (Stark, Bhutani 2016). Therefore, while the infant and the mother try to adapt to each other for successful breastfeeding, the treatment process increases breastfeeding difficulties and failure during the first postnatal week. The role and counseling of the infant's nurse are of great importance in breastfeeding of the newborn and the education of the family in neonatal jaundice. The first postnatal hours and days are the most critical times for ensuring the success of breastfeeding. Jaundice due to breastfeeding failure requires focused efforts for a program structured with breastfeeding education and special breastfeeding support. This support causes the role of nurses to become even more important.

Method: This is a randomized controlled experimental study. The data of the study will be collected from primiparous mothers who had normal delivery in the Gynecology and Obstetrics Department in Sakarya Maternity and Children's Hospital Campus affiliated to the Ministry of Health Sakarya University Training and Research Hospital between 01.08.2020-01.01.2021 and their infants until January 2021. The sample of the study was calculated in accordance with the intervention group selection criteria and by performing power analysis. Power analysis was performed using G*Power (v3.1.7) program in order to determine sample size. The effect range value was taken as 0.70 as the method used in cases where it is unknown how many units difference is significant between the groups. In cases where Type 1 error probability (α) was 0.05 (at a confidence level of 95%), at a power level of 80% and the effect range was 0.70, the study was planned with a total of 68 mothers, including 34 mothers women for each group. The mothers to be allocated to the study and control groups will be ensured to have similarity in terms of three factors (age, educational status, gender of the infants). The individuals will be allocated into groups by simple random sampling. The sample of the study will be randomly allocated into two groups: the intervention group will be supported for breastfeeding and the feeding of infants' with breast milk, and the other group, which was the control group, will be followed in routine care of the service. Single-blind (researchers are not blind) randomization will be provided since the mothers will be provided with support for breastfeeding and the feeding of infants' with breast milk by the researchers. The statistician was also blinded for the data analysis purpose. With regard to data collection tools, the "Mother Introductory Information Form" including socio-demographic characteristics of the family, the "Newborn Introductory Information Form" including characteristic features of the infants, the "Infant Nutrition Follow-up Form" for the follow-up of breast milk milked after breastfeeding, and the "Jaundice Follow-up Form" including the follow-up of infants who are hospitalized due to jaundice before/after discharge will be used. Mothers in the experimental group will be provided with breastfeeding support, and if required, the mother's both breasts will be milked by hand and the resulting breast milk will be collected in a container. After milking, the milk will be given to the infant with the help of a teaspoon. This practice will be shown to the mother and will be performed after each feeding during the hospital stay. Mothers will be told to perform this practice at home until the infant sucks effectively and strongly, and families will be called by phone daily. No intervention will be made to the control group. Bilirubin measurements of both groups will be performed with a transcutaneous bilirubin meter both before discharge from the hospital and at the end of week 1, and the values will be recorded. At the same time, the conditions of rehospitalization due to jaundice at the end of week 1 will be recorded. In the evaluation of data, statistical analyses will be performed using the SPSS package program. The Kolmogorov-Smirnov (K-S) test will be used for normality. In order to determine whether there is a difference in the dependent variables compared to independent variables, the independent group t-test will be used if the distribution is normal in independent variables with two options, and Mann Whitney-U test will be used if distribution is not normal. The results will be evaluated at a confidence level of 95% and at a level of significance of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* • Normal delivery of the mother

  * Mother being primiparous
  * Newborn being >38 GW
  * Having no multiple infants
  * Absence of congenital anomaly (craniofacial abnormality such as cleft palate, cleft lip, paralysis of facial muscles) in the newborn
  * No blood incompatibility between mother and father
  * Exclusive breastfeeding of the newborn
  * Non-contraindication of the mother's milk to her infant
  * Absence of the mother's diagnosed psychiatric story
  * Mother's openness to communication and cooperation
  * Mother's volunteering to participate in the study
  * Mother being literate
  * Mother's age above 18 years

Exclusion Criteria:

* • Separation of the mother and the infant due to any situation

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — breastfeeding mothers'
Enrollment: 68 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of bilirubin with a Transcutaneous bilirubinometer in the study and control groups | Change between the 1 day of discharge from hospital and the 7th day
  The device is suitable for use in newborn infants. The device measures by reader head's contact with the infant's forehead and by preventing user's possibility of making a mistake. The device shows the result on the LCD screen after 5 separate readings or has single and average measurement system. A value of above 5-7 mg/dl in the newborn is hyperbilirubinemia.

SECONDARY OUTCOMES:
hospitalization due to jaundice in the study and control groups | 7 days after discharge
  The study and control groups will be checked to see if they are hospitalized due to jaundice. Jaundice Follow-up Form created by the researchers includes questions status do hospitalizations

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Tabakoglu, MSc, Principal Investigator — Sakarya University; Vedat Cinar, MSc, Principal Investigator — Sakarya University; nursan cinar, professor, Study Director — Sakarya University; Sultan Peksen, Principal Investigator — Sakarya University Training and Research Hospital; özge Karakaya Suzan, MSc, Principal Investigator — Sakarya University
Locations (1):
- sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
typically after the end of the study

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/15231951/
- See also: Related Info — https://www.aafp.org/afp/2014/0601/p873.html